CLINICAL TRIAL: NCT04884984
Title: Pilot Study of the Safety and Efficacy of Anti-CLL1 Chimeric Antigen Receptor Engineered T-Cells in the Treatment of CLL1 Positive Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Anti-CLL1 CAR T-cell Therapy in CLL1 Positive Relapsed/Refractory Acute Myeloid Leukemia (AML)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UnicarTherapy2021001
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: CLL1; CART; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLL1 positive relapsed or refractory acute myeloid leukemia (Experimental)
  Interventions: Biological: anti-CLL1 CART

INTERVENTIONS:
Biological: anti-CLL1 CART — Split intravenous infusion of anti-CLL1 CAR T cells [dose escalating infusion of (5-20)x10^6 anti-CLL1 CAR T cells/kg].

SUMMARY:
This is a single center, open-label phase 1/2 study to evaluate the safety and efficacy of anti-CLL1 chimeric antigen receptor engineered T cell immunotherapy (CART) in the treatment of CLL1 positive relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
The patients will receive infusion of anti-CLL1 CAR T-cells to confirm the safety and efficacy of anti-CLL1 CAR T-cells in relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* CLL1 positive relapsed/refractory acute myeloid leukemia
* Age 6-65 years
* Left ventricular ejection fractions ≥ 0.5 by echocardiography
* Creatinine < 1.6 mg/dL
* Aspartate aminotransferase/aspartate aminotransferase < 3x upper limit of normal
* Total bilirubin <2.0 mg/dL
* Karnofsky performance status ≥ 60
* Expected survival time ≥ 3 months (according to investigator's judgement)

Exclusion Criteria:

* Patients are pregnant or lactating
* Uncontrolled active infection
* Class III/IV cardiovascular disability according to the New York Heart Association Classification
* Active hepatitis B or hepatitis C infection
* Patients with HIV infection
* Patients with history of seizure
* Active central nervous system leukemia

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)#Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)#All CR criteria except for residual neutropenia (<1.0x10^9/L) or thrombocytopenia (<100x10^9/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
overall survival (OS) | 2 years
  The date of enrollment to the date of death from any cause
Event-free survival (EFS) | 2 years
  Time from enrollment to the date of primary refractory disease, or relapse from CR or CRi, or death from any cause
Cumulative incidence of relapse(CIR) | 2 years
  Time from the date of achievement of a remission to the date of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China